CLINICAL TRIAL: NCT00945581
Title: Evaluation of AN777 on Elderly Subjects During Bed Rest and Recovery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK37
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Aged
Keywords: Healthy Elderly volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AN777 (Experimental): Powder twice a day
  Interventions: Other: Experimental Nutritional Powder Formula
- Placebo powder (Placebo Comparator): Powder twice a day
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: Experimental Nutritional Powder Formula — Powder twice a day
  Arms: AN777
Other: Placebo comparator — Powder twice a day
  Arms: Placebo powder

SUMMARY:
The primary objectives are to evaluate the effect of AN777 on muscle strength loss that occurs during bed rest, and to investigate whether AN777, in association with resistance training, will support muscle strength recovery following bed rest in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject (male or female) is > 60 to < 79 years of age.
* Subject has Body Mass Index (BMI)> 20 < 35.
* Subject is ambulatory with an SPPB score of > 9.
* Subject agrees to comply with prescribed activity level.

Exclusion Criteria:

* Subject has undergone major surgery, less than 4 weeks prior to enrollment in the study.
* Subject has stated active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix.
* Subject has stated history of diabetes or fasting glucose value > 126 mg/dL.
* Subject has stated presence of partial or full artificial limb.
* Subject has stated kidney disease or serum creatinine > 1.4 mg/dL.
* Subject has evidence of cardiovascular disease assessed during resting or exercise EKG.
* Subject has untreated hypothyroidism with TSH levels greater than 5.5 microUnits/ml.
* Subject has serum glutamate pyruvate transaminase (SGPT) levels greater than two times upper limit of laboratory-designated normal value.
* Subject has a history of allergy to any of the ingredients in the study products.
* Subject has an obstruction of the gastrointestinal tract precluding ingestion of the study product, inflammatory bowel disease, short bowel syndrome or other major gastrointestinal disease such as gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis.
* Subject has stated uncontrolled severe diarrhea, nausea or vomiting.

Subject is actively pursuing weight loss.

* Subject is currently taking medications/dietary supplements/substances that could modulate metabolism or weight in the opinion of the principal investigator or physician, e.g. progestational agents, steroids, growth hormone, dronabinol, marijuana, beta-hydroxyl-beta-methylbutyrate (HMB), free amino acid supplements, dietary supplements to aid weight loss. Exceptions for multi-vitamin/mineral supplement, inhaled steroids for asthma, topical or optical steroids and short-term use (less than two weeks) of Dexamethasone.
* Subject cannot refrain from smoking/discontinue the use of nicotine or tobacco.
* Subject has a stated history of Deep Vein Thrombosis (DVT) or a known hypercoaguable condition.
* Subject cannot discontinue current anticoagulant therapy.
* Subject has refractory anemia with hemoglobin value < 11.5 g/dL.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Lower extremity muscle strength changes after 10 days of bed rest, followed by changes after an 8-week recovery period. | 10 weeks

SECONDARY OUTCOMES:
Lower extremity lean body mass | 10 weeks
Muscle functionality | 10 weeks
Total lean mass | 10 weeks
physical activity levels | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Pereira, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626